CLINICAL TRIAL: NCT03979339
Title: Feasibility of a New Technology for Isolating Circulating Tumour Cells in Selected Cancer Patients and Healthy Volunteers
Brief Title: Feasibility of a New Technology for Isolating Circulating Tumour Cells
Acronym: CTC-SMMiL-E
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CTC-SMMiL-E-1901; 2019-A01187-50 (Other: ANSM)
Record Dates: First submitted 2019-05-27; First posted 2019-06-07 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: HER2-positive Metastatic Breast Cancer; Ovarian Cancer; Hormone-resistant Prostate Cancer; Circulating Tumor Cell
Keywords: Circulating Tumour Cells; Selected cancer patients; New technology
MeSH Terms: conditions — Ovarian Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- blood sample collection (Experimental): For all participants whatever the group Groups 0 and 4: Healthy volunteers Group1: Metastatic HER2-positive breast cancer Group 2: Advanced CA-125 positive ovarian cancer Group 3: Metastatic PSA-positive castrate-resistant prostate cancer Participants will receive the following interventions because they are enrolled in the study: blood sample collection of 32mL (4x8mL in EDTA tubes)
  Interventions: Procedure: Blood sample collection

INTERVENTIONS:
Procedure: Blood sample collection — A total volume of 32 ml of blood will be collected in each subject and separated in 4 10-mL EDTA vacutainer tubes EDTA tubes of 8 mL each.

SUMMARY:
This is a prospective interventional single-site research with a collection of biological samples.

The primary objective of the trial is to assess the ability of the "new technology" to isolating circulating tumor cells (CTC) in selected cancer patients.

Five groups will be constitued: at first the Group 0: Healthy volunteers included for the spike-in test; and then the four groups, Group1: Metastatic HER2-positive breast cancer; Group 2: Advanced CA-125 positive ovarian cancer; Group 3: Metastatic PSA-positive castrate-resistant prostate cancer; Group 4: Healthy volunteers included as control).

In each group, the percentage of cases with identified circulating tumor cells will be estimated.

DETAILED DESCRIPTION:
This is a prospective interventional single-site research with a collection of biological samples ("Recherche Impliquant la Personne Humaine de type 2" according to French legislation).

First, a cohort of 20 healthy volunteers (Group 0: Healthy volunteers included for the spike-in test) will be constituted for the spike-in-test.

Then, recruitment of the three groups of 14 patients each (Group1: Metastatic HER2-positive breast cancer; Group 2: Advanced CA-125 positive ovarian cancer; Group 3: Metastatic PSA-positive castrate-resistant prostate cancer) and the control group of 14 healthy volunteers (Group 4: Healthy volunteers included as control) will be done in parallel.

In each group, the percentage of cases with identified circulating tumor cells will be estimated. Success will be defined as follows: the new technique has isolated putative circulating cells that have been confirmed as tumor cells by the immuno-histochemistry approach.

Circulating tumor cells (CTC) will be identified as followed:

* Group 1 - putative circulating cells isolated by the new technique must be tested as HER-2 positive using Fluorescence In Situ Hybridization (FISH) to be regarded as true CTC
* Group 2 - putative circulating cells isolated by the new technique must be tested as CA 125-positive using immuno-histochemistry (IHC) to be regarded as true CTC
* Group 3 - putative circulating cells isolated by the new technique must be tested as PSA-positive using IHC to be regarded as true CTC For the healthy volunteers included as controls, if putative circulating cells are observed, these healthy volunteers will be tested against the three markers (HER2, CA-125 and PSA).

Failure will be defined as follows: the technique failed to identify circulating tumor cells, either due to a technical issue, or because there was no cell identified by the new technique, or lastly because the identified cells were negative by the standard FISH or IHC technique.

The different characteristics of these cells will be described: size, cytological characteristics, number, etc.

Secondary collected samples will be frozen, and new technique for isolation of CTC will be applied a second time to describe the impact of freezing to the capacity for isolating the CTC.

The primary objective of the trial is to assess the ability of the "new technology" to isolating circulating tumor cells (CTC) in selected cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Registered with a social security system
* Signed, IRB-approved written informed consent
* Belonging to one of the following group:
* Group 1 - HER-2 positive breast cancer, defined as followed: histologically-proven, HER-2 positive breast cancer, with metastasis (stage IV) requiring first-line treatment
* Group 2 - Advanced ovarian cancer, defined as followed: histologically-proven, stage III or IV ovarian cancer requiring first-line chemotherapy
* Group 3 - Metastatic prostate cancer, defined as followed: histologically-proven, stage IV, castrate-resistant prostate cancer requiring chemotherapy with docetaxel or treatment with 2nd generation hormonal therapy (e.g. enzalutamide or abiraterone)
* Groups 0 and 4 - Healthy volunteers defined as followed: No prior personal history of malignant disease

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2020-03-11 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of cases with identified circulating tumor cells. | within 24 hours after inclusion (blood sample collection)
  To assess the ability of the "new technology" to isolating circulating tumor cells (CTC) in selected cancer patients.
  In each group, the percentage of cases with identified circulating tumor cells will be estimated.
  Success: the technique has isolated putative circulating cells that have been confirmed as tumor cells by the immuno-histochemistry approach.
  Failure: the technique failed to identify circulating tumor cells, either due to a technical issue, or because there was no cell identified by the new technique, or lastly because the identified cells were negative by the standard FISH or IHC technique.
  To be regarded as true CTC, Putative circulating cells isolated by the new technique must be tested as:
  * HER-2 positive using Fluorescence In Situ Hybridization (FISH) (Group 1)
  * CA 125-positive using immuno-histochemistry (IHC) (Group 2)
  * PSA-positive using IHC (Group 3)

SECONDARY OUTCOMES:
Description of the isolated circulating cell | within 24 hours after inclusion (blood sample collection)
  Describe the different characteristics of these cells: size, cytological characteristics, number ...
  These informations will allow to characterize the isolated circulating cells.
Percentage of cases with identified circulating tumor cells after frozen storage | within 24 hours after inclusion (blood sample collection)
  To assess the ability of the new technology to isolating CTC
  As secondary collected, collected samples will be frozen, and new technique for isolation of CTC will be applied a second time to describe the impact of freezing to our capacity for isolating the CTC.
  In each group, the percentage of cases with identified circulating tumor cells will be estimated.
  To be regarded as true CTC, Putative circulating cells isolated by the new technique must be tested as:
  * HER-2 positive using Fluorescence In Situ Hybridization (FISH) (Group 1)
  * CA 125-positive using immuno-histochemistry (IHC) (Group 2)
  * PSA-positive using IHC (Group 3)

CONTACTS AND LOCATIONS:
Overall Officials: Emilie KACZMAREK, MD, Principal Investigator — Medical Oncology Department - Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bednarz-Knoll N, Alix-Panabieres C, Pantel K. Plasticity of disseminating cancer cells in patients with epithelial malignancies. Cancer Metastasis Rev. 2012 Dec;31(3-4):673-87. doi: 10.1007/s10555-012-9370-z. PMID 22733306
- [Background] Allard WJ, Matera J, Miller MC, Repollet M, Connelly MC, Rao C, Tibbe AG, Uhr JW, Terstappen LW. Tumor cells circulate in the peripheral blood of all major carcinomas but not in healthy subjects or patients with nonmalignant diseases. Clin Cancer Res. 2004 Oct 15;10(20):6897-904. doi: 10.1158/1078-0432.CCR-04-0378. PMID 15501967
- [Background] Cristofanilli M, Budd GT, Ellis MJ, Stopeck A, Matera J, Miller MC, Reuben JM, Doyle GV, Allard WJ, Terstappen LW, Hayes DF. Circulating tumor cells, disease progression, and survival in metastatic breast cancer. N Engl J Med. 2004 Aug 19;351(8):781-91. doi: 10.1056/NEJMoa040766. PMID 15317891
- [Background] Cristofanilli M, Hayes DF, Budd GT, Ellis MJ, Stopeck A, Reuben JM, Doyle GV, Matera J, Allard WJ, Miller MC, Fritsche HA, Hortobagyi GN, Terstappen LW. Circulating tumor cells: a novel prognostic factor for newly diagnosed metastatic breast cancer. J Clin Oncol. 2005 Mar 1;23(7):1420-30. doi: 10.1200/JCO.2005.08.140. PMID 15735118
- [Background] Riethdorf S, Fritsche H, Muller V, Rau T, Schindlbeck C, Rack B, Janni W, Coith C, Beck K, Janicke F, Jackson S, Gornet T, Cristofanilli M, Pantel K. Detection of circulating tumor cells in peripheral blood of patients with metastatic breast cancer: a validation study of the CellSearch system. Clin Cancer Res. 2007 Feb 1;13(3):920-8. doi: 10.1158/1078-0432.CCR-06-1695. PMID 17289886
- [Background] Yagata H, Nakamura S, Toi M, Bando H, Ohno S, Kataoka A. Evaluation of circulating tumor cells in patients with breast cancer: multi-institutional clinical trial in Japan. Int J Clin Oncol. 2008 Jun;13(3):252-6. doi: 10.1007/s10147-007-0748-9. Epub 2008 Jun 14. PMID 18553236
- [Background] Kurihara T, Itoi T, Sofuni A, Itokawa F, Tsuchiya T, Tsuji S, Ishii K, Ikeuchi N, Tsuchida A, Kasuya K, Kawai T, Sakai Y, Moriyasu F. Detection of circulating tumor cells in patients with pancreatic cancer: a preliminary result. J Hepatobiliary Pancreat Surg. 2008;15(2):189-95. doi: 10.1007/s00534-007-1250-5. Epub 2008 Apr 6. PMID 18392713
- [Background] Khoja L, Backen A, Sloane R, Menasce L, Ryder D, Krebs M, Board R, Clack G, Hughes A, Blackhall F, Valle JW, Dive C. A pilot study to explore circulating tumour cells in pancreatic cancer as a novel biomarker. Br J Cancer. 2012 Jan 31;106(3):508-16. doi: 10.1038/bjc.2011.545. Epub 2011 Dec 20. PMID 22187035
- [Background] Maheswaran S, Sequist LV, Nagrath S, Ulkus L, Brannigan B, Collura CV, Inserra E, Diederichs S, Iafrate AJ, Bell DW, Digumarthy S, Muzikansky A, Irimia D, Settleman J, Tompkins RG, Lynch TJ, Toner M, Haber DA. Detection of mutations in EGFR in circulating lung-cancer cells. N Engl J Med. 2008 Jul 24;359(4):366-77. doi: 10.1056/NEJMoa0800668. Epub 2008 Jul 2. PMID 18596266
- [Background] Nagrath S, Sequist LV, Maheswaran S, Bell DW, Irimia D, Ulkus L, Smith MR, Kwak EL, Digumarthy S, Muzikansky A, Ryan P, Balis UJ, Tompkins RG, Haber DA, Toner M. Isolation of rare circulating tumour cells in cancer patients by microchip technology. Nature. 2007 Dec 20;450(7173):1235-9. doi: 10.1038/nature06385. PMID 18097410
- [Background] Stott SL, Hsu CH, Tsukrov DI, Yu M, Miyamoto DT, Waltman BA, Rothenberg SM, Shah AM, Smas ME, Korir GK, Floyd FP Jr, Gilman AJ, Lord JB, Winokur D, Springer S, Irimia D, Nagrath S, Sequist LV, Lee RJ, Isselbacher KJ, Maheswaran S, Haber DA, Toner M. Isolation of circulating tumor cells using a microvortex-generating herringbone-chip. Proc Natl Acad Sci U S A. 2010 Oct 26;107(43):18392-7. doi: 10.1073/pnas.1012539107. Epub 2010 Oct 7. PMID 20930119
- [Background] Stott SL, Lee RJ, Nagrath S, Yu M, Miyamoto DT, Ulkus L, Inserra EJ, Ulman M, Springer S, Nakamura Z, Moore AL, Tsukrov DI, Kempner ME, Dahl DM, Wu CL, Iafrate AJ, Smith MR, Tompkins RG, Sequist LV, Toner M, Haber DA, Maheswaran S. Isolation and characterization of circulating tumor cells from patients with localized and metastatic prostate cancer. Sci Transl Med. 2010 Mar 31;2(25):25ra23. doi: 10.1126/scitranslmed.3000403. PMID 20424012
- [Background] Cen P, Ni X, Yang J, Graham DY, Li M. Circulating tumor cells in the diagnosis and management of pancreatic cancer. Biochim Biophys Acta. 2012 Dec;1826(2):350-6. doi: 10.1016/j.bbcan.2012.05.007. Epub 2012 Jun 7. PMID 22683404
- [Background] Soeth E, Grigoleit U, Moellmann B, Roder C, Schniewind B, Kremer B, Kalthoff H, Vogel I. Detection of tumor cell dissemination in pancreatic ductal carcinoma patients by CK 20 RT-PCR indicates poor survival. J Cancer Res Clin Oncol. 2005 Oct;131(10):669-76. doi: 10.1007/s00432-005-0008-1. Epub 2005 Sep 1. PMID 16136352
- [Background] Hoffmann K, Kerner C, Wilfert W, Mueller M, Thiery J, Hauss J, Witzigmann H. Detection of disseminated pancreatic cells by amplification of cytokeratin-19 with quantitative RT-PCR in blood, bone marrow and peritoneal lavage of pancreatic carcinoma patients. World J Gastroenterol. 2007 Jan 14;13(2):257-63. doi: 10.3748/wjg.v13.i2.257. PMID 17226905
- [Background] de Albuquerque A, Kubisch I, Breier G, Stamminger G, Fersis N, Eichler A, Kaul S, Stolzel U. Multimarker gene analysis of circulating tumor cells in pancreatic cancer patients: a feasibility study. Oncology. 2012;82(1):3-10. doi: 10.1159/000335479. Epub 2012 Jan 20. PMID 22270149
- [Background] Alix-Panabieres C, Pantel K. Circulating tumor cells: liquid biopsy of cancer. Clin Chem. 2013 Jan;59(1):110-8. doi: 10.1373/clinchem.2012.194258. Epub 2012 Sep 26. PMID 23014601
- [Background] Pantel K, Speicher MR. The biology of circulating tumor cells. Oncogene. 2016 Mar 10;35(10):1216-24. doi: 10.1038/onc.2015.192. Epub 2015 Jun 8. PMID 26050619
- [Background] Smerage JB, Barlow WE, Hortobagyi GN, Winer EP, Leyland-Jones B, Srkalovic G, Tejwani S, Schott AF, O'Rourke MA, Lew DL, Doyle GV, Gralow JR, Livingston RB, Hayes DF. Circulating tumor cells and response to chemotherapy in metastatic breast cancer: SWOG S0500. J Clin Oncol. 2014 Nov 1;32(31):3483-9. doi: 10.1200/JCO.2014.56.2561. Epub 2014 Jun 2. PMID 24888818
- [Background] Wan L, Pantel K, Kang Y. Tumor metastasis: moving new biological insights into the clinic. Nat Med. 2013 Nov;19(11):1450-64. doi: 10.1038/nm.3391. PMID 24202397
- [Background] Gorges TM, Kuske A, Rock K, Mauermann O, Muller V, Peine S, Verpoort K, Novosadova V, Kubista M, Riethdorf S, Pantel K. Accession of Tumor Heterogeneity by Multiplex Transcriptome Profiling of Single Circulating Tumor Cells. Clin Chem. 2016 Nov;62(11):1504-1515. doi: 10.1373/clinchem.2016.260299. Epub 2016 Sep 14. PMID 27630154
- [Background] Zhang Z, Shiratsuchi H, Palanisamy N, Nagrath S, Ramnath N. Expanded Circulating Tumor Cells from a Patient with ALK-Positive Lung Cancer Present with EML4-ALK Rearrangement Along with Resistance Mutation and Enable Drug Sensitivity Testing: A Case Study. J Thorac Oncol. 2017 Feb;12(2):397-402. doi: 10.1016/j.jtho.2016.07.027. Epub 2016 Aug 6. PMID 27507192
- [Background] Jordan NV, Bardia A, Wittner BS, Benes C, Ligorio M, Zheng Y, Yu M, Sundaresan TK, Licausi JA, Desai R, O'Keefe RM, Ebright RY, Boukhali M, Sil S, Onozato ML, Iafrate AJ, Kapur R, Sgroi D, Ting DT, Toner M, Ramaswamy S, Haas W, Maheswaran S, Haber DA. HER2 expression identifies dynamic functional states within circulating breast cancer cells. Nature. 2016 Sep 1;537(7618):102-106. doi: 10.1038/nature19328. Epub 2016 Aug 24. PMID 27556950
- [Background] van de Stolpe A, Pantel K, Sleijfer S, Terstappen LW, den Toonder JM. Circulating tumor cell isolation and diagnostics: toward routine clinical use. Cancer Res. 2011 Sep 15;71(18):5955-60. doi: 10.1158/0008-5472.CAN-11-1254. Epub 2011 Sep 6. PMID 21896640
- [Background] Gorges TM, Tinhofer I, Drosch M, Rose L, Zollner TM, Krahn T, von Ahsen O. Circulating tumour cells escape from EpCAM-based detection due to epithelial-to-mesenchymal transition. BMC Cancer. 2012 May 16;12:178. doi: 10.1186/1471-2407-12-178. PMID 22591372
- [Background] Vila A, Abal M, Muinelo-Romay L, Rodriguez-Abreu C, Rivas J, Lopez-Lopez R, Costa C. EGFR-Based Immunoisolation as a Recovery Target for Low-EpCAM CTC Subpopulation. PLoS One. 2016 Oct 6;11(10):e0163705. doi: 10.1371/journal.pone.0163705. eCollection 2016. PMID 27711186
- [Background] Mostert B, Kraan J, Bolt-de Vries J, van der Spoel P, Sieuwerts AM, Schutte M, Timmermans AM, Foekens R, Martens JW, Gratama JW, Foekens JA, Sleijfer S. Detection of circulating tumor cells in breast cancer may improve through enrichment with anti-CD146. Breast Cancer Res Treat. 2011 May;127(1):33-41. doi: 10.1007/s10549-010-0879-y. Epub 2010 Apr 9. PMID 20379845
- [Background] Alunni-Fabbroni M, Sandri MT. Circulating tumour cells in clinical practice: Methods of detection and possible characterization. Methods. 2010 Apr;50(4):289-97. doi: 10.1016/j.ymeth.2010.01.027. Epub 2010 Jan 29. PMID 20116432
- [Background] Lowes LE, Allan AL. Recent advances in the molecular characterization of circulating tumor cells. Cancers (Basel). 2014 Mar 13;6(1):595-624. doi: 10.3390/cancers6010595. PMID 24633084
- [Background] Vona G, Sabile A, Louha M, Sitruk V, Romana S, Schutze K, Capron F, Franco D, Pazzagli M, Vekemans M, Lacour B, Brechot C, Paterlini-Brechot P. Isolation by size of epithelial tumor cells : a new method for the immunomorphological and molecular characterization of circulatingtumor cells. Am J Pathol. 2000 Jan;156(1):57-63. doi: 10.1016/S0002-9440(10)64706-2. PMID 10623654
- [Background] Farace F, Massard C, Vimond N, Drusch F, Jacques N, Billiot F, Laplanche A, Chauchereau A, Lacroix L, Planchard D, Le Moulec S, Andre F, Fizazi K, Soria JC, Vielh P. A direct comparison of CellSearch and ISET for circulating tumour-cell detection in patients with metastatic carcinomas. Br J Cancer. 2011 Sep 6;105(6):847-53. doi: 10.1038/bjc.2011.294. Epub 2011 Aug 9. PMID 21829190
- [Background] Zheng S, Lin HK, Lu B, Williams A, Datar R, Cote RJ, Tai YC. 3D microfilter device for viable circulating tumor cell (CTC) enrichment from blood. Biomed Microdevices. 2011 Feb;13(1):203-13. doi: 10.1007/s10544-010-9485-3. PMID 20978853
- [Background] Karabacak NM, Spuhler PS, Fachin F, Lim EJ, Pai V, Ozkumur E, Martel JM, Kojic N, Smith K, Chen PI, Yang J, Hwang H, Morgan B, Trautwein J, Barber TA, Stott SL, Maheswaran S, Kapur R, Haber DA, Toner M. Microfluidic, marker-free isolation of circulating tumor cells from blood samples. Nat Protoc. 2014 Mar;9(3):694-710. doi: 10.1038/nprot.2014.044. Epub 2014 Feb 27. PMID 24577360
- [Background] Ozkumur E, Shah AM, Ciciliano JC, Emmink BL, Miyamoto DT, Brachtel E, Yu M, Chen PI, Morgan B, Trautwein J, Kimura A, Sengupta S, Stott SL, Karabacak NM, Barber TA, Walsh JR, Smith K, Spuhler PS, Sullivan JP, Lee RJ, Ting DT, Luo X, Shaw AT, Bardia A, Sequist LV, Louis DN, Maheswaran S, Kapur R, Haber DA, Toner M. Inertial focusing for tumor antigen-dependent and -independent sorting of rare circulating tumor cells. Sci Transl Med. 2013 Apr 3;5(179):179ra47. doi: 10.1126/scitranslmed.3005616. PMID 23552373
- [Background] Jaeger BAS, Neugebauer J, Andergassen U, Melcher C, Schochter F, Mouarrawy D, Ziemendorff G, Clemens M, V Abel E, Heinrich G, Schueller K, Schneeweiss A, Fasching P, Beckmann MW, Scholz C, Friedl TWP, Friese K, Pantel K, Fehm T, Janni W, Rack B. The HER2 phenotype of circulating tumor cells in HER2-positive early breast cancer: A translational research project of a prospective randomized phase III trial. PLoS One. 2017 Jun 6;12(6):e0173593. doi: 10.1371/journal.pone.0173593. eCollection 2017. PMID 28586395
- [Background] Zhang S, Li L, Wang T, Bian L, Hu H, Xu C, Liu B, Liu Y, Cristofanilli M, Jiang Z. Real-time HER2 status detected on circulating tumor cells predicts different outcomes of anti-HER2 therapy in histologically HER2-positive metastatic breast cancer patients. BMC Cancer. 2016 Jul 25;16:526. doi: 10.1186/s12885-016-2578-5. PMID 27456503
- [Background] Agelaki S, Kalykaki A, Markomanolaki H, Papadaki MA, Kallergi G, Hatzidaki D, Kalbakis K, Mavroudis D, Georgoulias V. Efficacy of Lapatinib in Therapy-Resistant HER2-Positive Circulating Tumor Cells in Metastatic Breast Cancer. PLoS One. 2015 Jun 17;10(6):e0123683. doi: 10.1371/journal.pone.0123683. eCollection 2015. PMID 26083256
- See also: Circulating tumor cells: potential markers of minimal residual disease in ovarian cancer? a study of the OVCAD consortium — https://www.ncbi.nlm.nih.gov/pubmed/29290959
- See also: The added value of circulating tumor cells examination in ovarian cancer staging — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4697683/
- See also: Vimentin and Ki67 expression in circulating tumour cells derived from castrate-resistant prostate cancer — https://www.ncbi.nlm.nih.gov/pubmed/26923772